CLINICAL TRIAL: NCT00004138
Title: The Utility of Positron Emission Tomography (PET) in Staging of Patients With Potentially Operable Non-Small Cell Lung Carcinoma
Brief Title: Positron Emission Tomography for Detecting Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z0050; CDR0000067368 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET scan + surgery (Experimental): Patients receive fludeoxyglucose F 18 (FDG) IV followed 45-60 minutes later by positron emission tomography (PET) imaging. Confirmatory studies, such as biopsy, fine needle aspiration, or other imaging studies are then conducted to confirm the PET findings.
  Patients with no mediastinal nodal or distant metastases identified by FDG-PET scan may undergo thoracotomy and pulmonary resection within 1 month of evaluation.
  Patients are followed at 5-6 months after surgery.
  Interventions: Procedure: positron emission tomography; Procedure: radionuclide imaging; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: positron emission tomography
Procedure: radionuclide imaging
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Imaging procedures, such as positron emission tomography (PET), may improve the ability to detect the extent of non-small cell lung cancer.

PURPOSE: Diagnostic trial to study the effectiveness of PET for detecting lesions in patients who have newly diagnosed stage I, stage II, or stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective: To ascertain whether FDG-PET scanning can detect lesions that would preclude pulmonary resection in patients found to be surgical candidates by standard imaging procedures.

Secondary Objectives: To use the data collected to generate hypotheses to be used in future studies, such as which types of previously undetected lesions FDG-PET is best able to identify.

Patients receive fludeoxyglucose F 18 (FDG) IV followed 45-60 minutes later by positron emission tomography (PET) imaging. Confirmatory studies, such as biopsy, fine needle aspiration, or other imaging studies are then conducted to confirm the PET findings.

Patients with no mediastinal nodal or distant metastases identified by FDG-PET scan may undergo thoracotomy and pulmonary resection within 1 month of evaluation.

Patients are followed at 5-6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥ 18 years of age.
2. a) Patient must have histologically or cytologically confirmed, newly diagnosed, untreated, single lesion bronchogenic NSCLC (adenocarcinoma, non-lobar/non- diffuse bronchioloalveolor cell carcinoma, large cell carcinoma, or squamous cell carcinoma). OR b) Patient is eligible based upon mediastinal node histology diagnosed by transbronchial biopsy, and if a separate ipsilateral lung lesion is clearly evident on radiographs, biopsy of the lung tumor is not required for this patient. OR c) Patient may be eligible without histologic or cytologic proof if;

   * The patient is strongly suspected to have primary bronchogenic carcinoma (e.g., heavy smoker with a new peripheral mass with typical appearance of lung cancer on chest radiograph although bronchoscopy and/or fine needle aspiration is nondiagnostic), and
   * The tumor is clinically resectable, and
   * An exploratory thoracotomy is planned.
3. Patient must be medically fit for surgical staging procedures following the thoracic surgeon's evaluation of general medical fitness.
4. Patient must be a candidate for resection of the clinical stage I, II, or IIIa lesion.
5. Patient must be able to tolerate PET, (i.e., not claustrophobic and able to lie supine for 1.5 hrs).
6. A signed and dated written informed consent must be obtained from the patient or the patient's legally acceptable representative prior to study participation.
7. Female patient of childbearing potential must have a negative serum or urine pregnancy test, 72 hours prior to FDG-PET.

   * NOTE: This is in order to avoid unnecessary fetal radiation exposure and because the use of furosemide is contraindicated in pregnancy.
8. Patient must complete the following standard staging procedures 60 days prior to registration.

   * CT scan of the chest and upper abdomen (include adrenals) with contrast
   * NOTE: Non-contrast CT scan may be used for patients with a peripheral suspicious nodule and no evidence of hilar or mediastinal adenopathy or invasion of central structures. All other lesions require IV contrast.
   * Bone scan
   * CT scan of the brain with and without contrast or MRI of brain
9. A cancer survivor is eligible provided that ALL the following criteria are met and documented:

   * the patient has undergone potentially curative therapy for all prior malignancies, and
   * there has been no evidence of any prior malignancies for at least five years (except for completely resected cervical or non-melanoma skin cancer), and
   * the patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Exclusion Criteria:

1. Patient has had a prior PET scan for evaluation of their NSCLC.
2. Patient has evidence of stage IIIB or IV disease confirmed by diagnostic imaging such as chest X-ray, CT chest, CT abdomen, CT brain or MRI brain, and bone scan.
3. Patient has uncontrolled diabetes mellitus, as evidenced by a fasting blood glucose value >200 mg/dL, within 12 hours of PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 1999-09; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with negative findings from FDG-PET scan | Up to 1 month post-FDG-PET scan

SECONDARY OUTCOMES:
Proportion of false-positive lesions found by FDG-PET | Up to 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn E. Reed, MD, Study Chair — Medical University of South Carolina
Locations (23):
- United States (23):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Veterans Affairs Medical Center - Iowa City, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Westmoreland Hospital, Greensburg, Pennsylvania
  - Jameson Memorial Hospital, New Castle, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Kozower BD, Meyers BF, Reed CE, Jones DR, Decker PA, Putnam JB Jr. Does positron emission tomography prevent nontherapeutic pulmonary resections for clinical stage IA lung cancer? Ann Thorac Surg. 2008 Apr;85(4):1166-9; discussion 1169-70. doi: 10.1016/j.athoracsur.2008.01.018. PMID 18355490
- [Result] Reed CE, Harpole DH, Posther KE, Woolson SL, Downey RJ, Meyers BF, Heelan RT, MacApinlac HA, Jung SH, Silvestri GA, Siegel BA, Rusch VW; American College of Surgeons Oncology Group Z0050 trial. Results of the American College of Surgeons Oncology Group Z0050 trial: the utility of positron emission tomography in staging potentially operable non-small cell lung cancer. J Thorac Cardiovasc Surg. 2003 Dec;126(6):1943-51. doi: 10.1016/j.jtcvs.2003.07.030. PMID 14688710